CLINICAL TRIAL: NCT01957969
Title: French Post-Inscription Study on Sacral Neuromodulation in the Treatment of Fecal Incontinence
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Collaborators: Medtronic France SAS (Industry); Medtronic MCRI (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1.05.8004
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Principal Population: Patients who undergo a definitive neuro-stimulator implantation.
  Interventions: Device: Sacral Nerve Stimulation
- Annex Population: Patients who do not respond to the temporary test for the neurostimulator implantation
  Interventions: Device: Sacral Nerve Stimulation

INTERVENTIONS:
Device: Sacral Nerve Stimulation
  Other Names: INTERSTIM

SUMMARY:
The aim of this observational study is to evaluate the utilization in the clinical practice, effectiveness, explantation and re-intervention rate, complications and adverse events of InterStim system in patients indicated to Sacral Neuromodulation therapy for fecal incontinence.

This study will provide additional data about safety and effectiveness of the usage of InterStim system in fecal incontinence environment and at the same time will confirm that results from clinical trials can be transposed to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to sign the Data Release Form stating the non opposition to the study conduct;
* Patient able to understand information given by the investigator in terms of data collection and publication;
* At least 18 years old or older.
* Patient indicated to sacral neuromodulation testing with InterStim® system.

Exclusion Criteria:

* Replacement of an existing sacral neuromodulation system (implanted before inclusion period) without any evidence of benefits during a testing period.
* Patient unwilling to comply to data collection and publication rules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French subjects affected by fecal incontinence, indicated to sacral neuromodulation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2013-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of implanted patients with a reduction of at least 50% of incontinence episodes per week, compared to baseline. | 6 months (4-8 months)
  The primary objective will evaluate the proportion of implanted patients that do not experience any serious adverse event or serious adverse device effect at 4-8 months of follow-up and show a reduction of at least 50% of incontinence episodes per week at the same timeframe, compared to baseline.

SECONDARY OUTCOMES:
Reduction of incontinence episodes per week | 12 months (9-15 months)
Reduction of evacuations per week | 6 months (4-8 months) and 12 months (9-15 months)
Reduction of urgency episodes per week | 6 months (4-8 months) and 12 months (9-15 months)
Retention delay | 3 months (1-4 months), 6 months (5-8 months), 12 months (9-15 months)
Complications and Adverse Events | 3 months (1-4 months), 6 months (5-8 months), 12 months (9-15 months)
Fecal Incontinence severity | 3 months (1-4 months), 6 months (5-8 months), 12 months (9-15 months)
Quality of Life | 3 months (1-4 months), 6 months (5-8 months), 12 months (9-15 months)
Patient Satisfaction | 6 months (5-8 months) and 12 months (9-15 months)

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - CHU Estaing, Clermont-Ferrand
  - CHU Grenoble - Hôpital Michallon, Grenoble
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - CHU Dupuytren, Limoges
  - Hopital Edouard Herriot, Lyon
  - APM Hopital Nord, Marseille
  - CHU Nantes - Hotel Dieu, Nantes
  - GH Diaconesses Croix St Simon, Paris
  - Hôpital Saint Joseph, Paris
  - CHU La Milétrie, Poitiers
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU Charles Nicolle, Rouen
  - Polyclinique Pays Basque Sud, Saint-Jean-de-Luz
  - CHU Hautepierre, Strasbourg
  - CHU Toulouse - Hotel Dieu PURPAN, Toulouse
  - Clinique St Jean du Languedoc, Toulouse

REFERENCES:
- [Background] Matzel KE, Kamm MA, Stosser M, Baeten CG, Christiansen J, Madoff R, Mellgren A, Nicholls RJ, Rius J, Rosen H. Sacral spinal nerve stimulation for faecal incontinence: multicentre study. Lancet. 2004 Apr 17;363(9417):1270-6. doi: 10.1016/S0140-6736(04)15999-0. PMID 15094271
- [Background] Jarrett ME, Varma JS, Duthie GS, Nicholls RJ, Kamm MA. Sacral nerve stimulation for faecal incontinence in the UK. Br J Surg. 2004 Jun;91(6):755-61. doi: 10.1002/bjs.4545. PMID 15164447
- [Background] Uludag O, Koch SM, van Gemert WG, Dejong CH, Baeten CG. Sacral neuromodulation in patients with fecal incontinence: a single-center study. Dis Colon Rectum. 2004 Aug;47(8):1350-7. doi: 10.1007/s10350-004-0589-9. PMID 15484349
- [Background] Altomare DF, Rinaldi M, Lobascio P, Marino F, Giuliani RT, Cuccia F. Factors affecting the outcome of temporary sacral nerve stimulation for faecal incontinence. The value of the new tined lead electrode. Colorectal Dis. 2011 Feb;13(2):198-202. doi: 10.1111/j.1463-1318.2009.02088.x. PMID 19863601
- [Background] Mellgren A, Wexner SD, Coller JA, Devroede G, Lerew DR, Madoff RD, Hull T; SNS Study Group. Long-term efficacy and safety of sacral nerve stimulation for fecal incontinence. Dis Colon Rectum. 2011 Sep;54(9):1065-75. doi: 10.1097/DCR.0b013e31822155e9. PMID 21825885
- [Background] Altomare DF, Ratto C, Ganio E, Lolli P, Masin A, Villani RD. Long-term outcome of sacral nerve stimulation for fecal incontinence. Dis Colon Rectum. 2009 Jan;52(1):11-7. doi: 10.1007/DCR.0b013e3181974444. PMID 19273950
- [Background] Wexner SD, Coller JA, Devroede G, Hull T, McCallum R, Chan M, Ayscue JM, Shobeiri AS, Margolin D, England M, Kaufman H, Snape WJ, Mutlu E, Chua H, Pettit P, Nagle D, Madoff RD, Lerew DR, Mellgren A. Sacral nerve stimulation for fecal incontinence: results of a 120-patient prospective multicenter study. Ann Surg. 2010 Mar;251(3):441-9. doi: 10.1097/SLA.0b013e3181cf8ed0. PMID 20160636
- [Background] Tjandra JJ, Chan MK, Yeh CH, Murray-Green C. Sacral nerve stimulation is more effective than optimal medical therapy for severe fecal incontinence: a randomized, controlled study. Dis Colon Rectum. 2008 May;51(5):494-502. doi: 10.1007/s10350-007-9103-5. Epub 2008 Feb 16. PMID 18278532
- [Background] Leroi AM, Parc Y, Lehur PA, Mion F, Barth X, Rullier E, Bresler L, Portier G, Michot F; Study Group. Efficacy of sacral nerve stimulation for fecal incontinence: results of a multicenter double-blind crossover study. Ann Surg. 2005 Nov;242(5):662-9. doi: 10.1097/01.sla.0000186281.09475.db. PMID 16244539
- [Background] Tan E, Ngo NT, Darzi A, Shenouda M, Tekkis PP. Meta-analysis: sacral nerve stimulation versus conservative therapy in the treatment of faecal incontinence. Int J Colorectal Dis. 2011 Mar;26(3):275-94. doi: 10.1007/s00384-010-1119-y. Epub 2011 Jan 29. PMID 21279370
- [Background] Matzel KE, Lux P, Heuer S, Besendorfer M, Zhang W. Sacral nerve stimulation for faecal incontinence: long-term outcome. Colorectal Dis. 2009 Jul;11(6):636-41. doi: 10.1111/j.1463-1318.2008.01673.x. Epub 2008 Aug 21. PMID 18727721
- [Derived] Meurette G, Siproudhis L, Leroi AM, Damon H, Urs Josef Keller D, Faucheron JL; French Faecal Registry Study Group. Sacral neuromodulation with the InterStim system for faecal incontinence: results from a prospective French multicentre observational study. Colorectal Dis. 2021 Jun;23(6):1463-1473. doi: 10.1111/codi.15507. Epub 2021 Mar 12. PMID 33387373